CLINICAL TRIAL: NCT01456078
Title: A Multicenter Phase II-Study Evaluating Efficacy and Safety of 177Lu-DOTA-TATE Based on Kidney-Dosimetry in Patients With Disseminated Neuroendocrine Tumors
Brief Title: A Multicenter Study Evaluating Efficacy and Safety of 177Lu-DOTA-TATE Based on Kidney-Dosimetry in Patients With Disseminated Neuroendocrine Tumors
Acronym: ILUMINET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number: 2011-000240-16
Record Dates: First submitted 2011-10-07; First posted 2011-10-20 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Neuroendocrine Tumors; Liver Metastases
Keywords: Neuroendocrine tumor; Liver metastases; 177Lu-DOTA-TATE; Safety; Kidney dosimetry; Dose escalation; Neuroendocrine tumors, with liver metastases.
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 177Lu-DOTA-TATE (Experimental)
  Interventions: Drug: 177Lu-DOTA-TATE

INTERVENTIONS:
Drug: 177Lu-DOTA-TATE — 177Lu-DOTA-TATE given as intravenous infusion given during 3-5 treatments. Evaluation is performed after every single cycle. Further more, evaluation is made after last cycle, and delivered cumulative dose to kidneys should be 27 Gy.
  Patients with stable disease or partial response, and without pronounced toxicity will continue treatment to a step 2, where additional 3-5 treatment cycles are given, with a cumulative dose to kidneys to 40 Gy.

SUMMARY:
By improved kidney dosimetry including biological effective dose and taking into account potential risk factors (especially for kidney toxicity), it might be possible to give an optimal and personalized treatment with 177Lu-DOTA-TATE to the patient with metastatic neuroendocrine tumor.

ELIGIBILITY:
Inclusion Criteria:

Step 1:

* ECOG 0-2
* Histologically verified neuroendocrine tumors with a Ki67 of at least 20 % or at least 20 mitoses/high power fields. If the tissue on which this determination is based is several years old, the investigator should consider the option of acquiring a new determination, especially if the behaviour of the tumor has changed since diagnosis
* Metastatic disease where complete resection is not considered possible or feasible
* Measurable disease
* Radiological disease progression during the last 14 months
* The largest metastases should have an uptake of 111In-octreotide that is greater than the uptake in the liver by planar scintigraphy. Metastases that are small, or located centrally, can be evaluated by SPECT to enable a correct estimation of the relative uptake. The majority of the tumor burden must demonstrate an increased uptake for lutetium-treatment to be considered
* Stable dose of somatostatin analogue for the past 3 months
* Estimated survival more than 6 months
* ANC more than 1.5 x 10 9/L
* Bilirubin less than 1.5 x upper limit of normal
* GFR more than 50 ml/min.
* Signed written informed concent

Step 2:

* Continues to fulfill all of the inclusion criteria, and none of the exclusion criteria, from step 1
* A maintained GFR (less than 40 % decrease compared to baseline AND GFR more than 50 ml/min)
* The treatment in step 1 have been administered with a maximal interval of 12 weeks
* Age under 70 years

Exclusion Criteria:

Step 1:

* Performance Status ECOG 3-4
* Proliferation index (Ki67) more than 20 % or more than 20 mitoses/hpf
* Loco-regional treatment during the last 3 months involving all of the measurable lesions
* Chemotherapy during the last 3 months, or longer if persisting toxicity exists. Earlier treatment with mTORi or TKI is permitted
* Other concommitant nephrotoxic treatment
* Modifications of the somatostatine dose in the last 3 months
* Serious heart disease
* Previous radiotherapy including more than 25 % of active bone marrow volume
* Pregnancy and lactation
* Extensive liver metastases (more than 50 % of liver volume)
* Symptomatic CNS metastases requiring corticosteroid treatment
* Ongoing treatment with interferon. This treatment should be suspended a minimum of 4 weeks before treatment with 177Lu-DOTA-TATE, or longer if there is persisting signs of toxicity
* Patients who have another metastatic tumor diagnosis

Step 2:

* Progressive disease since start of study treatment
* Organ toxicity grade 3-4 during step 1
* Serious hematological toxicity during previous treatment cycles (ANC less than 0.5 x 10 9 or platelets less than 50.0 x 10 9)
* Longstanding diabetes (more than 8 years). Patients with a well-controlled diabetes with a history of less than 8 years and a blood pressure less than 130/80 and no albuminuria (albumin/creatinine index)can be included
* Hypertension, i.e. more than 160/90 (for diabetics more than 130/80). Antihypertensive pharmacological treatment is permitted as long as there is no manifest albuminuria
* Previous liver embolisation
* Previous chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Objective tumor response after a cumulative kidney biologically effective dose (BED) of 27 +/- 2 Gy | 3 months after completed step 1

SECONDARY OUTCOMES:
Objective tumor response after receiving a cumulative BED to the kidneys of 40 +/- 2 Gy as per RECIST v 1.1 | 3 months after completing step 2 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tennvall, MD, PhD, Principal Investigator — Department of Oncology, Lund University Hospital
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Department of Oncology, Gothenburg
  - Department of Oncology, Lund University Hospital, Lund

REFERENCES:
- [Derived] Sundlov A, Gleisner KS, Tennvall J, Ljungberg M, Warfvinge CF, Holgersson K, Hallqvist A, Bernhardt P, Svensson J. Phase II trial demonstrates the efficacy and safety of individualized, dosimetry-based 177Lu-DOTATATE treatment of NET patients. Eur J Nucl Med Mol Imaging. 2022 Sep;49(11):3830-3840. doi: 10.1007/s00259-022-05786-w. Epub 2022 Apr 22. PMID 35451612